CLINICAL TRIAL: NCT00740961
Title: The Vulnerable Elders Survey Study of Older Cancer Patients
Brief Title: Older Patients With Newly Diagnosed Breast Cancer or Colon Cancer
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE8Y07
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Colorectal Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; cognitive/functional effects; breast cancer; colon cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Colonic Neoplasms | interventions — Neoadjuvant Therapy; Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 13mls of blood will be drawn at each of the three time-points for testing for biologic correlates of frailty (pre study, mid-study and post-study).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with cancer: Patients ≥ 65 years with new stage I-III breast or colon cancer seeking care. Patients will be matched on baseline scores, age and sex. Patients will be age and sex matched due to the known relation between inflammatory markers and demographic characteristics39,40, and will be matched on baseline VES scores to ensure similar baseline VES-13 scores between groups and which will then allow us to then assess effect of cancer treatment on outcomes.
  Interventions: Behavioral: compliance monitoring; Drug: systemic chemotherapy; Other: medical chart review; Other: study of socioeconomic and demographic variables; Other: survey administration; Procedure: cognitive assessment; Procedure: psychosocial assessment and care
- Patients without cancer: non-cancer patients, seeking care at out-patient clinics
  Interventions: Behavioral: compliance monitoring; Other: medical chart review; Other: study of socioeconomic and demographic variables; Other: survey administration; Procedure: cognitive assessment; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: compliance monitoring — Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.
Drug: systemic chemotherapy — Learning about changes over time in older patients' ability to function after receiving chemotherapy for breast or colon cancer
  Groups: Patients with cancer
Other: medical chart review — A limited review of medical records for the sole purpose of evaluating patients for study eligibility will be undertaken by the research team.
Other: study of socioeconomic and demographic variables — Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.
Other: survey administration — Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.
Procedure: cognitive assessment — Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.
Procedure: psychosocial assessment and care — Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.

SUMMARY:
RATIONALE: Learning about changes over time in older patients' ability to function after receiving chemotherapy for breast or colon cancer may help doctors learn about the long-term effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying older patients with newly diagnosed breast cancer or colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the correlation between the Vulnerable Elders Survey (VES-13) and the battery of Comprehensive Geriatric Assessment tools among breast and colon cancer patients, 65 years and older, in an outpatient setting.
* Assess and compare the abilities of the VES-13 and the battery of Comprehensive Geriatric Assessment tools to predict chemotherapy adherence among these patients.
* Examine the validity of the VES-13 screening tool to identify increased risk of death from all causes at one year after initial VES-13 screening in these patients.
* Examine the validity of the VES-13 screening tool to identify increased risk of functional decline at one year after initial VES-13 screening in these patients.

OUTLINE: Patients complete the Vulnerable Elders Survey (VES-13) and a Comprehensive Geriatric Assessment at baseline and 12 months later. Variables collected include sociodemographics; cognitive, nutritional, psychosocial, and emotional status; tumor characteristics; therapy; and mortality.

Patients are followed for 1 year for chemotherapy adherence and survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast or colon cancer

  * Newly diagnosed disease
  * Any stage disease
* Undergoing treatment at the Ireland Cancer Center, University Hospitals Case Medical Center Site
* Scheduled to start a new chemotherapy regimen (objective II only)
* Not concurrently enrolled in a GEM trial (objectives II, III, and IV)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Understands English
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Diseases Characteristics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary Care clinic
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of impaired domains on Comprehensive Geriatric Assessment (CGA) | at baseline and 12 months later.
Chemotherapy adherence as measured by dose reduction, dose delay, and grade 3-5 toxicities | Patients are followed for 1 year for chemotherapy adherence and survival.
Vulnerable Elders Survey scores | at baseline and 12 months later.
Functional decline | at baseline and 12 months later.
Time to death | Patients are followed for 1 year for chemotherapy adherence and survival.

SECONDARY OUTCOMES:
Scores of individual battery of tools included in the CGA | at baseline and 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, MD, MSC, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-LUICC, Mentor, Ohio
  - UH-Chagrin Highlands, Orange, Ohio
  - UH-Green Road, South Euclid, Ohio
  - UH-Westlake, Westlake, Ohio